CLINICAL TRIAL: NCT02075879
Title: The Effects of a Nurse-led Case Management Programme on Home Exercise Training for Haemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Susan Ka Yee Chow, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSEARS20121105002
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Kidney Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse-led interviewing (Experimental): Participants in experimental arm received the in-center exercise training (20 minutes) before hemodialysis sessions weekly for 6 weeks and were instructed to perform exercise at home. They were additionally instructed to start walking or brisk walking at low duration and gradually progress to a maximum of 30 minutes daily per week. To facilitate exercise progression, the nurse case managers discussed exercise benefits, explored exercise barriers and developed mutual goals with patients. The nurse motivated them and checked the exercise behaviors to ensure adherence to the recommended exercise regime. The nurse case managers interviewed the patients weekly for six weeks and biweekly for another six weeks.
  Interventions: Behavioral: Nurse-led interviewing
- Brief group exercise (Active Comparator): Participants received the in-center exercise training (20 minutes) before hemodialysis sessions weekly for 6 weeks and were instructed to perform exercise at home. The in-center training was conducted by the researcher with a group of four-to six participants focusing on flexibility and strengthening exercise only.
  Interventions: Other: Brief group exercise

INTERVENTIONS:
Behavioral: Nurse-led interviewing — Participants in experimental arm received regular face-to-face interviews during dialysis sessions conducted by the designated case managers every week for 6 weeks and biweekly for another 6 weeks.
  Arms: Nurse-led interviewing
Other: Brief group exercise — Participants in this arm only participated in the brief in-center exercise training. They received usual care from the nurse without the interviews and mutual goals developed.
  Arms: Brief group exercise

SUMMARY:
The purpose of this study is to examine the effects of a nurse-led case management programme on home exercise training for haemodialysis patients. We hypothesised that: a. There is no significant difference in physical functioning between participants receiving the nurse-led home exercise training programme and those receiving the comparison care. b. There is no difference in depression between participants receiving the nurse-led home exercise training programme and those receiving the comparison care. c. There is no difference in quality of life and health perception between participants receiving the nurse-led home exercise training programme and those receiving the comparison care. d. There is no difference in physical activity levels between participants receiving the nurse-led home exercise training programme and those receiving the comparison care. e. There is no difference in perceived benefits and barriers of exercise between participants receiving the nurse-led home exercise training programme and those receiving the comparison care.

The study was a randomized controlled trial conducted in two haemodialysis units of two tertiary hospitals in Nanjing, China. Participants were randomly assigned to either study group or comparison group. Participants in both groups received the in-center exercise training (20 minutes) before haemodialysis sessions weekly for 6 weeks and were instructed to perform exercise at home. The in-center training was focused on flexibility and strengthening exercise. Patients were encouraged to have cardiovascular exercises at home which will improve their cardiovascular conditions and endurance. The list of cardiovascular exercise included brisk walking, bicycling, jogging. Participants in the study group were instructed to start walking or brisk walking at low duration and gradually progress to a maximum of 30 minutes daily per week. To facilitate exercise progression, the nurse case managers discussed exercise benefits, explored exercise barriers and developed mutual goals with patients. The nurse motivated them and checked the exercise behaviors to ensure adherence to the recommended exercise regime. The nurse case managers interviewed the study group patients weekly for six weeks and biweekly for another six weeks. Participants in the comparison group only participated in the in-center exercise training. The comparison group patients received usual care from the nurse without the interviews and mutual goals developed.

DETAILED DESCRIPTION:
The duration of interventions was 12 weeks. In-center exercise training sessions were available for all participants once a week for 6 weeks. Each session lasted about 20 minutes. Participants were instructed to perform flexibility and strength exercise in centres prior to the haemodialysis session. The researcher performed exercises with the participants and emphasised the importance of self-monitoring during the sessions. Symptoms (such as chest pain, dyspnea, dizziness, and leg cramps) and vital signs (blood pressure, heart rate, and pulse) were checked before exercise and monitored during the entire exercise session. Participants were instructed to self-monitor exercise intensity. The exercise programme was pause immediately if the patient was feeling short of breath, chest pain or pressure, irregular heartbeats, leg cramps, dizziness or lightheadedness, blurring of vision, or any discomfort.

Intervention group During the study period, participants in the intervention group received additional face-to-face interviews conducted by the designated case managers every week for six weeks and biweekly for another six weeks. During interviews, patients were instructed to start aerobic exercise, such as walking, jogging, cycling, or brisk walking at home at low duration and gradually progress to a maximum of 30 minutes daily per week. Apart from aerobic exercise, patients were recommended to perform strength exercises twice a week and flexibility exercises for every day. The key elements of the interview included: 1) assessment of patients' knowledge and exercise behaviour; examining patients' attitudes and feelings about being physical activity; 2) explore patients' barriers to exercise and perceived benefits; 3) patient education on the benefits of exercise if needed; 4) development of mutual goals in an exercise plan; 5) explain the purpose of a recording exercise log and instruction in correct way to keep an exercise diary; 6) discuss the available supports and resources that could motivate patients to initiate and maintain exercise, e.g., centre-based exercise programme, support from family members, health care providers, peer patients, and so forth.

In the follow-up interviews, case managers reviewed the exercise log with participants, discussed unpleasant experiences related to exercise, exercise progress, and provided encouragement. According to the progress participants made, the exercise goals and plan were renewed or revised. Referrals were made as needed.

Comparison group Participants in the comparison group were advised to participate in the in-centre exercise training programme which was available before haemodialysis sessions once a week for different shifts of patients. The training session lasted about 20 minutes and only flexibility and strength training were provided. During the training sessions, patients were advised to increase their daily activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis for >3 months;
* Age > 18 years;
* Kt/V (dialysis adequacy) >1.2;
* Hemoglobin level > 8g/dl;
* Ambulatory without assistance ;
* Able to communicate in Chinese;
* Able to and willing to provide consent.

Exclusion Criteria:

* Unstable physical conditions or severe musculoskeletal diseases that might hinder exercise training;
* Severe hearing impairment;
* Diagnosed with mental diseases;
* Meeting or exceeding the exercise recommendation.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in walking speed on the 10-meter walking test at week 6 and change from baseline in walking speed on 10-meter walking test at week 12 | Baseline, Week 6, and Week 12

SECONDARY OUTCOMES:
Change from baseline in time in completing the 10-repetition sit-to-stand test (10-STS) at week 6, and change from baseline in time in completing 10-STS at week 12 | Baseline, Week 6, and Week 12
Change from baseline in perceived exercise benefits and barriers on the Dialysis Patient-perceived Exercise Benefits and Barriers Scale (DPEBBS) at week 6 and change from baseline in the DPEBBS score at week 12 | Baseline, Week 6, and Week 12
Change from baseline in health-related quality of life on the Kidney Disease Quality of Life Questionnaire (KDQOL-36) at week 6, and change from baseline in KDQOL-36 score at week 12 | Baseline, Week 6, and Week 12
Change from baseline in depressive symptoms on the Beck Depression Inventory (BDI) at week 6, and change from baseline in BDI score at week 12 | Baseline, Week 6, and Week 12
Change from baseline in self-perceived health in the first item in the Kidney Disease Quality of Life Questionnaire at week 6, and change from baseline in self-perceived health score at week 12 | Baseline, Week 6, and Week 12
Change from week 6 in physical activity levels measured by exercise log at week 12 | Week 6 and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Susan KY Chow, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (2):
- China (2):
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The Second Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Tao X, Chow SK, Wong FK. A nurse-led case management program on home exercise training for hemodialysis patients: A randomized controlled trial. Int J Nurs Stud. 2015 Jun;52(6):1029-41. doi: 10.1016/j.ijnurstu.2015.03.013. Epub 2015 Mar 26. PMID 25840898